CLINICAL TRIAL: NCT01077661
Title: An Open Label, Multi-centre, Non-interventional Post-marketing Surveillance (PMS) to Monitor the Safety and Effectiveness of Nebilet Administered in Korean Patients According to the Prescribing Information
Brief Title: Regulatory Nebilet PMS
Acronym: Nebilet PMS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113554
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Hypertension; Heart Failure
Keywords: Nebivolol; PMS (post-marketing surveillance)
MeSH Terms: conditions — Hypertension; Heart Failure | interventions — Nebivolol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients administrated Nebivolol: There is only one group. This group includes patients administrated Nebivolol
  Interventions: Drug: Nebivolol

INTERVENTIONS:
Drug: Nebivolol — patients administrated Nebivolol according to the prescribing information

SUMMARY:
An open label, multi-centre, non-interventional post-marketing surveillance (PMS) to monitor the safety and effectiveness of Nebivolol administered in Korean patients according to the prescribing information

DETAILED DESCRIPTION:
An open label, multi-centre, non-interventional post-marketing surveillance (PMS) to monitor the safety and effectiveness of Nebivolol administered in Korean patients according to the prescribing information

Nebivolol will be administered to Hypertension or Chronic heart failure (CHF) patients as described the prescribing information of Nebivolol by physician's decision.

ELIGIBILITY:
All subjects must satisfy the following criteria at PMS entry according to KFDA PMS regulation:

* Subjects with indication in the prescribing information
* Subjects administrated Nebivolol by physician's decision
* Subjects with no contraindication according to the prescribing information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients administrated Nebivolol at the site
Sampling Method: Probability Sample
Enrollment: 743 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events after Nebivolol administration | 3months, 6months

SECONDARY OUTCOMES:
Occurrence of unexpected or serious adverse event after Nebivolol administration and effectiveness of Occurrence of unexpected or serious adverse event after Nebivolol administration and effectiveness of Nebivolol | 3 months, 6months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea